CLINICAL TRIAL: NCT04957914
Title: Effects of LY3209590 on Frequency and Severity of Hypoglycaemia Under Conditions of Increased Hypoglycaemic Risk Compared to Insulin Glargine in Participants With Type 2 Diabetes Mellitus
Brief Title: A Study of LY3209590 on Low Blood Sugar in Participants With Type 2 Diabetes Mellitus
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Basic Science
Other Study IDs: 16936; I8H-MC-BDCI (Other: Eli Lilly and Company); 2019-003537-42 (EudraCT Number)
Record Dates: First submitted 2021-07-08; First posted 2021-07-12 (Actual); Last update posted 2022-11-16 (Actual); Status verified 2022-11-01

CONDITIONS: Type 2 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Insulin Glargine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Insulin Glargine (Period 1) (Active Comparator): Insulin glargine administered subcutaneously (SC).
  Interventions: Drug: Insulin Glargine
- LY3209590 (Period 2) (Experimental): LY3209590 administered SC.
  Interventions: Drug: LY3209590

INTERVENTIONS:
Drug: Insulin Glargine — Administered SC
  Arms: Insulin Glargine (Period 1)
Drug: LY3209590 — Administered SC
  Arms: LY3209590 (Period 2)

SUMMARY:
The main purpose of this study is to evaluate the effect of study drug known as LY3209590 compared to insulin glargine administered in participants with type 2 diabetes mellitus (T2DM). Side effects and tolerability will be documented. The study will last almost six months and 21 visits for each participant including screening period.

ELIGIBILITY:
Inclusion Criteria:

* Have been diagnosed with Type 2 Diabetes Mellitus (T2DM) for at least 1 year prior to screening
* Body mass index (BMI) of 18.5 to 40.0 kilograms per meter squared (kg/m²)
* Be treated for T2DM with stable dose of metformin, a stable dose of a dipeptidyl peptidase-4 (DPP-4) inhibitor with or without metformin, or a stable dose of a glucagon-like peptide-1 (GLP-1) receptor agonist with or without metformin for at least 3 months prior to screening

Exclusion Criteria:

* Have an abnormality in the 12-lead ECG
* Have a supine blood pressure at screening
* Have alanine aminotransferase (ALT) or aspartate aminotransferase (AST) >2.5x upper limit of normal (ULN)
* Have a history of or current cardiovascular, respiratory, hepatic, renal, gastrointestinal, endocrine (except T2DM and controlled thyroid disease), haematological, or neurological disorders
* Are receiving chronic (lasting longer than 14 consecutive days) systemic or inhaled glucocorticoid therapy
* Have an average weekly alcohol intake

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2021-07-14 (Actual); Primary Completion 2022-10-17 (Actual); Study Completion 2022-10-17 (Actual)

PRIMARY OUTCOMES:
Incidence of Documented Hypoglycemia | Baseline through Day 186
  Incidence of Documented Hypoglycemia

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (1):
- Profil Institut für Stoffwechselforschung, Neuss, North Rhine-Westphalia, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Heise T, Andersen G, Pratt EJ, Leohr J, Fukuda T, Wang Q, Kazda C, Bue-Valleskey JM, Bergenstal RM. Frequency and Severity of Hypoglycemia Under Conditions of Increased Hypoglycemic Risk with Insulin Efsitora Alfa Versus Insulin Glargine Treatment in Participants with Type 2 Diabetes. Diabetes Ther. 2024 Aug;15(8):1785-1797. doi: 10.1007/s13300-024-01605-7. Epub 2024 Jun 22. PMID 38907935